CLINICAL TRIAL: NCT06825975
Title: A Phase II Single-Arm Clinical Study to Explore the Efficacy and Safety of Hyperbaric Oxygen in the Neoadjuvant Treatment of Triple-Negative and HER2+ Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, PhD, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-1118-02
Record Dates: First submitted 2025-01-21; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancers
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyperbaric Oxygen group (Experimental): Patients who meet the inclusion criteria will be enrolled and given hyperbaric oxygen intervention, with a minimum of 5 times hyperbaric oxygen treatments per chemotherapy cycle, one per day for 60-90 minutes, for a total of 30-40 hyperbaric oxygen treatments (100% oxygen at a pressure of 2.0 ATA).
  Interventions: Device: Hyperbaric oxygen treatment

INTERVENTIONS:
Device: Hyperbaric oxygen treatment — Patients who meet the inclusion criteria will be enrolled and given hyperbaric oxygen intervention, with a minimum of 5 hyperbaric oxygen treatments per chemotherapy cycle, one per day for 60-90 minutes, for a total of 30-40 hyperbaric oxygen treatments (100% oxygen at a pressure of 2.0 ATA).

SUMMARY:
The goal of the study is to explore the efficacy and safety of hyperbaric oxygen therapy in the neoadjuvant treatment of triple-negative and HER2+ breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study process, participate in the study voluntarily, and sign the informed consent form.
2. have an initial histopathologically confirmed diagnosis of unilateral primary invasive breast cancer, excluding occult breast cancer, inflammatory breast cancer and eczema-like carcinoma
3. aged ≥ 18 years and ≤ 60 years, female
4. patients who meet the inclusion criteria of neoadjuvant therapy to receive neoadjuvant therapy for breast cancer (patients with locally advanced breast cancer (AJCC Stage III, except T3N1M0) or operable but not in breast-conserving or axillary-sparing condition (Stage IIA-IIB and T3N1M0), or patients with a certain tumour load of HER2-positive or TNBC with clinical lymph node positivity, or patients with a tumour size of 2cm and above). or tumour size 2cm and above).
5. ECOG performance status 0-1.
6. LVEF ≥ 55%
7. Adequate bone marrow functional reserve: white blood cell count ≥3.0 x 109/L, neutrophil count ≥1.5 x 109/L; platelet count ≥100 x 109/L; haemoglobin ≥90 g/L;
8. AST, ALT ≤ 2.5 times the upper limit of normal value, alkaline phosphatase ≤ 2.5 times the upper limit of normal value, total bilirubin ≤ 1.5 times the upper limit of normal value; serum creatinine ≤ 1.5 times the upper limit of normal value
9. For non-menopausal or non-surgically sterilised female patients: consent to contraception during treatment and for at least 7 months after the last dose of the study treatment

   -

Exclusion Criteria:

1. Contraindication to hyperbaric oxygen therapy: untreated pneumothorax. Concurrent use of disulfiram. concomitant administration of anti-tumour drugs such as bleomycin, cisplatin, adriamycin concomitant administration of antineoplastic drugs such as bleomycin, cisplatin, adriamycin. Premature and/or low body mass neonates. Lung disease (severe chronic obstructive pulmonary disease). Diseases of the lungs (severe chronic obstructive airway disease, herpetic lung disease, acute or chronic lung infections, uncontrolled asthma, uncontrolled diarrhoea). controlled asthma, untreated pneumothorax), history of previous middle ear surgery, middle ear disease (eustachian tube Dysfunction of the eustachian tube, recurrent episodes of vertigo), ocular disease (retinal detachment).
2. previous hyperbaric oxygen therapy.
3. distant metastases, including lymph node metastases to the contralateral breast and mediastinum.
4. other malignant tumours within the last two years, except for radically treated basal or squamous cell carcinoma of the skin or CIS of the cervix. Tumour.
5. pregnancy or lactation
6. uncontrolled hypertension, cardiac, hepatic, renal related disease or other medical or psychiatric conditions.
7. major surgical procedure unrelated to breast cancer within 4 weeks prior to randomisation, or the patient has not fully recovered from such procedure; or has not fully recovered from such surgical intervention.
8. serious or uncontrolled infections that may interfere with study treatment or assessment of study results, including but not limited to Serious or uncontrolled infections that may interfere with study treatment or the evaluation of study results, including but not limited to active hepatitis virus infection, human immunodeficiency virus (HIV) antibody positivity, and pulmonary infections.
9. recent history of thromboembolism and taking full dose anticoagulant medication.
10. any other condition that, in the opinion of the investigator, makes the patient unsuitable for participation in the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 348 (Estimated)
Dates: Start 2025-02-12 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR rate after hyperbaric oxygen combined with neoadjuvant therapy in breast cancer patients | After completion of standard cycle of neoadjuvant therapy (through study completion, an average of half a year)

SECONDARY OUTCOMES:
The Miller and payne classification | After completion of standard cycle of neoadjuvant therapy (through study completion, an average of half a year)
RCB 0/1 rate | After completion of standard cycle of neoadjuvant therapy (through study completion, an average of half a year)
  RCB (Residual Cancer Burden) is a commonly used metric to assess the extent of residual tumor burden after neoadjuvant therapy, such as chemotherapy, radiation therapy, or targeted therapy.
  RCB 0: Complete response (CR) - No visible residual tumor, complete disappearance of the tumor.
  RCB I: Minimal residual disease - Only a small amount of residual tumor remains, with limited tumor volume and few lymph node metastases.
  RCB II: Moderate residual disease - Moderate degree of tumor residual is present.
  RCB III: Extensive residual disease - A large amount of residual tumor remains, often with more lymph node metastases.
RECIST criteria | After completion of the first cycle of neoadjuvant therapy (at about 1 month), After completion of standard cycle of neoadjuvant therapy (through study completion, an average of half a year)
Life quality (EORTC QLQ C-30、EORTC QLQ BR-23 questionnaire) | At the time of patient enrolment, Each cycle of chemotherapy (8cycle, each cycle is 3 weeks) , Day before surgery, 3 months after surgery.
Side effects of hyperbaric oxygen therapy | during the hyperbaric oxygen therapy (up to half a year)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | through study completion ( an average of half a year)
the Tumor immune microenvironment of the Hyperbaric Oxygen Therapy and neoadjuvant therapy | the time when the patient enrollment, at the end of the first cycle of neoadjuvant therapy (at about the first month) , surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, China